CLINICAL TRIAL: NCT07242300
Title: A Phase III Clinical Study to Evaluate the Efficacy and Safety of Recombinant Botulinum Toxin Type A (Eveotox) in Adult Patients With Upper Limb Spasticity
Brief Title: Efficacy and Safety of Recombinant Botulinum Toxin Type A (Eveotox) for Injection in the Treatment of Adult Upper Limb Spasticity .
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: JHM BioPharma (Tonghua) Co. , Ltd. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JHM03-CT302
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Upper Limb Spasticity (ULS)
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): Eveotox will be administered in double-blind fashion at cycle 1 followed by up to 3 open-label cycles of Eveotox.
  Interventions: Drug: Recombinant Botulinum Toxin Type A for injection
- Placebo-Controlled Group (Placebo Comparator): Placebo will be administered in double-blind fashion during treatment cycle 1 only, followed by up to 3 cycles of Eveotox.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant Botulinum Toxin Type A for injection — Recombinant Botulinum Toxin Type A for injection
  Arms: Treatment Group
Drug: Placebo — Placebo will be administered in double-blind fashion during treatment cycle 1 only
  Arms: Placebo-Controlled Group

SUMMARY:
This is a phase III clinical study to evaluate the efficacy and safety of recombinant botulinum toxin type A（Eveotox）in adult patients with upper limb spasticity. The purpose of this study was to observe efficacy and safety of Eveotox compared with placebo in adult patients with upper limb spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 80 years of age inclusive, at the time of signing the informed consent
* Participants with stable post-stroke Spasticity (ULS) for at least 3 months
* Participants with Modified Ashworth Scale (MAS) score of at least 2 at elbow flexor or wrist flexor or finger flexor
* Participants with DAS score of at least 2 on the Principal Target of Treatment (PTT) (one of four functional domains: dressing, hygiene, limb position and pain)
* Participants who have been stable for at least 1 month prior to study entry in terms of oral antispasticity

Exclusion Criteria:

* Previous use of any botulinum toxin within 6 months prior to screening, or plan to use any botulinum toxin during the study.
* History of alcohol or drug abuse.
* Known allergy or hypersensitivity to any component of the study products.
* History of epilepsy
* Known or suspected to be HIV positive, serologically positive for syphilis, or active hepatitis B or C
* Any medical condition that may put the participant at increased risk for botulinum toxin type A use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | Within 4 weeks
  Change from baseline at week 4 for primary targeted muscle group on the MAS(Modified Ashworth Scale).

SECONDARY OUTCOMES:
Secondary Outcome Measure | Within 52 weeks
  Incidence of adverse events and drug-related adverse events during the study.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Yangzhi Affiliated Rehabilitation Hospital of Tongji University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No